CLINICAL TRIAL: NCT00477958
Title: Determining the Utility of an Assessment Tool for Older Patients With Cancer
Brief Title: Assessment Tool for Older Patients With Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 06170; P30CA033572 (NIH); CHNMC-06170; MSKCC-06034; CDR0000540332 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cognitive/Functional Effects; Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cognitive/functional effects; psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Geriatric Assessment Tool (Experimental)
  Interventions: Other: questionnaire administration; Procedure: cognitive assessment; Procedure: psychosocial assessment and care

INTERVENTIONS:
Other: questionnaire administration — Questionnaire administered prior to chemotherapy and within 30 days of completion of chemotherapy.
Procedure: cognitive assessment — Cognitive assessment to be obtained prior to chemotherapy and within 30 days of completion of chemotherapy.
Procedure: psychosocial assessment and care — Psychosocial assessment and care to be obtained prior to chemotherapy and within 30 days of completion of chemotherapy.

SUMMARY:
RATIONALE: A study that assesses the ability of older patients to think, learn, remember, make judgments, and carry out daily activities may help doctors plan treatment for older patients with cancer.

PURPOSE: This clinical trial is studying an assessment tool in older patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether a geriatric assessment tool can predict toxicity to chemotherapy, defined as grade 3 or 4 toxicity, hospitalization, dose delay or reduction, or discontinuation of chemotherapy due to toxicity, in elderly patients with cancer.

Secondary

* Explore the longitudinal impact of cancer and chemotherapy treatment on geriatric assessment parameters.

OUTLINE: Patients undergo assessments of functional status using the Timed Up and Go Assessment (measures physical mobility) and Karnofsky Physician-Rated Performance Rating Scale; and cognition using the Blessed Orientation-Memory-Concentration Test. These assessments are performed by healthcare personnel. Body mass index and the percentage of unintentional weight loss and the number of falls in the past 6 months are also assessed.

Patients also complete the following self-administered questionnaires: Instrumental Activities of Daily Living (measures level of functioning and need for services); Activities of Daily Living (measures higher levels of physical functioning); Karnofsky Self-Reported Performance Rating Scale (related to survival and clinically significant illness); Physical Health Section of the Older American Resources and Services Questionnaire (measures comorbidity and the impact on daily activities); Hospital Anxiety and Depression Scale; Medical Outcomes Study (MOS) Social Activity Limitations Measure (measures the impact of cancer on patients' social functioning); and MOS Social Support Survey Emotional/Information and Tangible Subscales (measures perceived availability of social support).

Patients then begin planned chemotherapy.

After completion of chemotherapy (or a maximum of 12 months from study entry), patients undergo assessments and complete self-administered questionnaires as described above.

PROJECTED ACCRUAL: A total of 750 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed cancer

  * Receiving chemotherapy for either adjuvant treatment or metastatic disease prior to beginning a new chemotherapy regimen

PATIENT CHARACTERISTICS:

* Must be able to understand English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior enrollment in this trial
* No concurrent enrollment on a phase I clinical trial

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1062 (Actual)
Dates: Start 2006-12-19 (Actual); Primary Completion 2015-07-27 (Actual); Study Completion 2026-03-13 (Estimated)

PRIMARY OUTCOMES:
Ability to predict toxicity to chemotherapy, defined as grade 3-4 toxicity, hospitalization, dose delay or reduction, or discontinuation of chemotherapy due to toxicity, as measured by a geriatric assessment tool | Prior to chemotherapy and within 30 days of completion of chemotherapy.

SECONDARY OUTCOMES:
Longitudinal impact of cancer and chemotherapy treatment on geriatric assessment parameters | Prior to chemotherapy and within 30 days of completion of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dale William, MD, Principal Investigator — City of Hope Medical Center
Locations (8):
- United States (8):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Medical Center, Duarte, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio